CLINICAL TRIAL: NCT04277182
Title: Effect of Topical Turkish Propolis Application on Burn Healing in Experimental Burn Model
Brief Title: Effect of Propolis Application on Burn Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, ESRA ARDAHAN AKGUL, Research Assistant, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-048
Record Dates: First submitted 2020-02-17; First posted 2020-02-20 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Burns; Burn Wound
Keywords: Burn; Burn wound; Propolis; Wound healing
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: * 1st. group: It will be considered as a control group and rats will not be treated.
  * 2nd. group: Vehicle group, Propolis vehicle will be applied to rats for 21 days.
  * 3rd. group: Silver Sulfadiazine group, 1% Silver Sulfadiazine will be applied topically to rats for 21 days.
  * 4th. group: Nitrafurozon group, 0.2% Nitrafurozon will be applied topically for 21 days.
  * 5th. group: 10% Propolis group, 10% Propolis will be applied topically for 21 days.
  * 6th. group: 15% Propolis group, 15% Propolis will be applied topically for 21 days.
Who Masked: Outcomes Assessor
Masking Description: the researcher who will analyze the primary outcome of the study will not know which group of animals the samples were taken from.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control group (Placebo Comparator): It will be accepted as the control group and 4 experimental burn wounds will be created on the back of the rats in the group and no treatment will be given.
  Interventions: Biological: burn wound dressing
- 1% Silver Sulfadiazine (Active Comparator): 4 experimental burn wounds will be created on the back of the rats in the group and dressing with 1% Silver Sulfadiazine will be done on the back of the rats every day for 21 days.
  Interventions: Biological: burn wound dressing
- %0.2 Nitrafurozon (Active Comparator): 4 experimental burn wounds will be created on the back of the rats in the group and dressing with %0.2 Nitrafurozon will be done on the back of the rats every day for 21 days.
  Interventions: Biological: burn wound dressing
- 10% Propolis (Experimental): 4 experimental burn wounds will be created on the back of the rats in the group and dressing with 10% Propolis will be done on the back of the rats every day for 21 days.
  Interventions: Biological: burn wound dressing
- 15% Propolis (Experimental): 4 experimental burn wounds will be created on the back of the rats in the group and dressing with 15% Propolis will be done on the back of the rats every day for 21 days.
  Interventions: Biological: burn wound dressing
- Propolis vehicle (Active Comparator): 4 experimental burn wounds will be created on the back of the rats in the group and dressing with Propolis vehicle will be done on the back of the rats every day for 21 days.
  Interventions: Biological: burn wound dressing

INTERVENTIONS:
Biological: burn wound dressing — 1. st. group: It will be considered as a control group and rats will not be treated.
  2. nd. group: Vehicle group, Propolis vehicle will be applied topically to rats for 21 days.
  3. rd group: Silver Sulfadiazine group, 1% Silver Sulfadiazine will be applied topically to rats for 21 days.
  4. th. group: Nitrafurozon group, 0.2% Nitrafurozon will be applied topically for 21 days.
  5. th. group: 10% Propolis group, 10% Propolis will be applied topically for 21 days.
  6. th. group: 15% Propolis group, 15% Propolis will be applied topically for 21 days.

SUMMARY:
This experimental study will be carried out at Ege University Laboratory Animals Application and Research Center to identify the efficacy of 10% propolis and 15% propolis on wound healing in a second-degree superficial burn wound.

In the study, 36 adult (8-12 week old) Wistar-Albino rats with a weight of 200-300 grams will be used in each group. Each group will include 6 rats. Stratified randomization will be used to randomize rats according to their gender and weight. After randomization, a burnt area will be created on the back of the rats and dressings will be made every day.

Following the creation of the burn, biopsy samples will be taken on the 3rd, 7th, 14th and 21st days and at the light microscopic level; bulla, erythema, oedema, burn depth, inflammatory cell infiltration, necrosis, ulceration, angiogenesis, neovascularization, fibroblast proliferation, collagenization, epithelization, fibrosis, the number of hair follicles and damage to the skin attachments.

In the immunohistochemical examination of biopsy samples, samples will be taken for the evaluation of superoxide dismutase, malondialdehyde, myeloperoxidase in the evaluation of the tumour necrosis factor-alpha, interleukin-1β and oxidative stress in the EBB period in order to evaluate the acute phase reactants. Fungal and gram staining will be done in order to determine the pathogen reproduction in biopsy samples taken on the 3rd and 7th day. Masson trichrome in order to detect fibrosis in biopsy samples taken on the 14th and 21st day; Hydroxyproline examination will be examined in order to evaluate collagen formation.

ELIGIBILITY:
Inclusion Criteria:

* adult (8-12 weeks)
* 200-300 grams
* Wistar-Albino rat
* with 4 second-degree superficial contact burn are at its back.

Exclusion Criteria:

* the death of the rat in the research process

Ages: 8 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
wound size | 21 days
  photos will be taken every day to determine the wound size
bulla | 3rd day of the research
  examination of the skin at the light microscopic level. Bulla will be considered as present or absent.
bulla | 7th day of the research
  examination of the skin at the light microscopic level. Bulla will be considered as present or absent.
bulla | 14th day of the research
  examination of the skin at the light microscopic level. Bulla will be considered as present or absent.
bulla | 21st day day of the research
  examination of the skin at the light microscopic level. Erythemawill be considered as present or absent.
edema | 3rd day of the research
  examination of the skin at the light microscopic level. Edema will be considered as present or absent.
edema | 7th day of the research
  examination of the skin at the light microscopic level. Edema will be considered as present or absent.
edema | 14th day of the research
  examination of the skin at the light microscopic level. Edema will be considered as present or absent.
edema | 21st day of the research
  examination of the skin at the light microscopic level. Edema will be considered as present or absent.
inflammatory cell infiltration | 3rd day of the research
  examination of the skin at the light microscopic level. Inflammatory cell infiltration will be considered as present or absent.
inflammatory cell infiltration | 7th day of the research
  examination of the skin at the light microscopic level. Inflammatory cell infiltration will be considered as present or absent.
inflammatory cell infiltration | 14th day of the research
  examination of the skin at the light microscopic level. Inflammatory cell infiltration will be considered as present or absent.
inflammatory cell infiltration | 21st day of the research
  examination of the skin at the light microscopic level. Inflammatory cell infiltration will be considered as present or absent.
necrosis | 3rd day of the research
  examination of the skin at the light microscopic level. Necrosis will be considered as present or absent.
necrosis | 7th day of the research
  examination of the skin at the light microscopic level. Necrosis will be considered as present or absent.
necrosis | 14th day of the research
  examination of the skin at the light microscopic level. Necrosis will be considered as present or absent.
necrosis | 21st day of the research
  examination of the skin at the light microscopic level. Necrosis will be considered as present or absent.
ulceration | 3rd day of the research
  examination of the skin at the light microscopic level. Ulceration will be considered as present or absent.
ulceration | 7th day of the research
  examination of the skin at the light microscopic level. Ulceration will be considered as present or absent.
ulceration | 14th day of the research
  examination of the skin at the light microscopic level. Ulceration will be considered as present or absent.
ulceration | 21st day of the research
  examination of the skin at the light microscopic level. Ulceration will be considered as present or absent.
angiogenesis | 3rd day of the research
  examination of the skin at the light microscopic level. Angiogenesis will be considered as present or absent.
angiogenesis | 7th day of the research
  examination of the skin at the light microscopic level. Angiogenesis will be considered as present or absent.
angiogenesis | 14th day of the research
  examination of the skin at the light microscopic level. Angiogenesis will be considered as present or absent.
angiogenesis | 21st day of the research
  examination of the skin at the light microscopic level. Angiogenesis will be considered as present or absent.
fibroblast proliferation | 3rd day of the research
  examination of the skin at the light microscopic level. Fibroblast proliferation will be considered as present or absent.
fibroblast proliferation | 7th day of the research
  examination of the skin at the light microscopic level. Fibroblast proliferation will be considered as present or absent.
fibroblast proliferation | 14th day of the research
  examination of the skin at the light microscopic level. Fibroblast proliferation will be considered as present or absent.
fibroblast proliferation | 21st day of the research
  examination of the skin at the light microscopic level. Fibroblast proliferation will be considered as present or absent.
epithelization | 3rd day of the research
  examination of the skin at the light microscopic level. Epithelization will be considered as present or absent.
epithelization | 7th day of the research
  examination of the skin at the light microscopic level. Epithelization will be considered as present or absent.
epithelization | 14th day of the research
  examination of the skin at the light microscopic level. Epithelization will be considered as present or absent.
epithelization | 21st day of the research
  examination of the skin at the light microscopic level. Epithelization will be considered as present or absent.
collagenization | 3rd day of the research
  examination of the skin at the light microscopic level. Collagenization will be considered as present or absent.
collagenization | 7th day of the research
  examination of the skin at the light microscopic level. Collagenization will be considered as present or absent.
collagenization | 14th day of the research
  examination of the skin at the light microscopic level. Collagenization will be considered as present or absent.
collagenization | 21st day of the research
  examination of the skin at the light microscopic level. Collagenization will be considered as present or absent.
microorganism colonization | 3rd day of the research
  examination of the skin at the light microscopic level. Colonization will be considered as present or absent.
microorganism colonization | 7th day of the research
  examination of the skin at the light microscopic level. Colonization will be considered as present or absent.
microorganism colonization | 14th day of the research
  examination of the skin at the light microscopic level. Colonization will be considered as present or absent.
microorganism colonization | 21st day of the research
  examination of the skin at the light microscopic level. Colonization will be considered as present or absent.

CONTACTS AND LOCATIONS:
Overall Officials: Figen Yardımcı, Study Director — Ege University
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
the study's data is planned to be published and shared in a scientific paper